CLINICAL TRIAL: NCT02631993
Title: Photochemotherapy of Acute Graft-versus-host Disease (aGVHD) of the Skin - is Graft-versus-leukemia Preserved in Patients Transplanted for Acute Leukemia?
Brief Title: Photochemotherapy and Graft-versus-leukemia in Acute-leukemia
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Nicolas Feldreich, M.D., Karolinska University Hospital
Other Study IDs: TIM Photochem 2
Record Dates: First submitted 2015-09-08; First posted 2015-12-16 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: ALL; AML; Acute GVHD; Tumor Immunity
Keywords: Psoralen; UVA; Time-to-treatment; GVL
MeSH Terms: interventions — Photochemotherapy; Ficusin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Photochemotherapy — Oral 8-Methoxypsoralene (8-MOP), (0.4-0.8 mg/kg), are given 1.5-2 hours before phototherapy. Ultraviolet light type A (UVA, 320-400 nm) is administered in a Waldmann UV1000 supine unit through 26 100-W fluorescent PUVA lamps (Waldmann F85), if needed, UVA is given in a half body unit with 15 100-W PUVA-lamps (Waldmann F85), (Waldmann UV3003K), (Waldmann, Villingen-Schwenningen, Germany). Eye protection is applied during 24 h after oral 8-MOP and the genital area are shielded in males during therapy.The UVA is initiated at 0.2-1.5 J/cm2 and is amplified by 0.25-0.5 J/cm2 after two treatments if photo toxicity is absent. PUVA is given to the patients 3-5 times each week.
  Other Names: Psoralen and Ultraviolet light Type A (PUVA)

SUMMARY:
Cure of leukemia after hematopoietic stem cell transplantation (HSCT) is sustained by the anti-leukemic effect of the grafted cells (graft-versus-leukemia (GVL)). However, it is not known whether the tumor-immunity is affected by photochemotherapy (psoralene photosensitization and ultraviolet light radiation) administered to attenuate graft-versus host disease (GVHD).

The present study aim to investigate what happens to the GVL after photochemotherapy of aGVHD in a predominantly retrospective setting with 10-years follow-up after HSCT

DETAILED DESCRIPTION:
This is a 10-year follow-up of patients with Acute-myeloid-leukemia (AML) or acute-lymphatic-leukemia (ALL). AML is diagnosed by the French-American-British criteria (FAB-criteria) and ALL is separated into chief forms by immunohistological methods. All patients underwent myeloablative Hematopoietic Stem Cell Transplantation (HSCT) between 1985 and 2005 at the center for allogeneic stem cell transplantation (CAST) at Karolinska University Hospital. All patient receive GVHD-prophylaxis.

The risk for relapse after HSCT is graded into low-risk if the disease is in first complete remission before HSCT, all other disease states are classified as high-risk.

Eligible patients received photochemotherapy (Ultraviolet radiation type A on skin photosensitized by oral 8-methoxypsoralen) for acute graft-versus-host disease (GVHD within 100-days after HSCT). Photochemotherapy may be given as primary or later aGVHD therapy. Patients with aGVHD after booster doses of stem-cells or donor-lymphocyte-infusions are not included.

Additional treatment are registered where present. Methotrexate is not considered as an additional GVHD treatment as intravenous methotrexate a part of the governing GVHD prophylaxis and as the effects of methotrexate as a secondary aGVHD treatment is weak.

At the start, the end, at maximum and up until two weeks after end of PUVA-therapy the GVHD is diagnosed in accordance with Glucksberg and indexed by CIBMTR.

Relapse is diagnosed when leukemic cells is present extra medullary or with a bone marrow biopsy with ≥ 30% blasts. Early relapse is diagnosed when the medulla contain 5 - 30% blasts

The primary outcome is GVL i.e. abscence of relapse in malignant disease or minimal residual disease (MRD) i.e. threatening relapse in malignant disease demanding donor lymphocyte infusion (DLI).

Primary predictor: Time-to-treatment by photochemotherapy at day 0 - 7 vs. start at day 8 ≤ of aGVHD.

Continuous secondary predictor: Time-to-treatment by photochemotherapy as a continuous variable (days after start of aGVHD).

Binary secondary predictors: Risk (Low/High), Sibling donor-recipient (Yes/No), Mismatched related (Yes/No), Unrelated donor (Yes/No), (Male recipients of female grafts (Yes/No), T-cell depletion or Anti-Thymocyte Globulin (Yes/No).

Categorical secondary predictors: AGVHD organ disease stage and disease grade; Skin (+, ++, +++, ++++), Liver (+, ++, +++, ++++), Gastro-intestinal (+, ++, +++, ++++), Center for International Blood and Marrow Transplant Research CIBMTR index (A, B, C, D) respectively.

Statistical analysis:

Cox proportional Hazards ratio is used to conduct a univariate data analysis of all adequate variables in patient characteristics and disease towards the primary outcome. In the analysis, death, DLI or retransplantation due to graft-failure was treated as a competing event. The primary predictor (binary) and all binary or categorical covariates identified from the patient and disease characteristics are to be included in a multivariate forward regression analysis, controlled for with backward regression based on the log-likelihood method. P=0.05 is considered as significant and p=0.10 as a trend. StatSoft, Inc. (2013). STATISTICA (data analysis software system), version 12. www.statsoft.com. are used for statistical computation.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients received photochemotherapy (Ultraviolet radiation type A on skin photosensitized by oral 8-methoxypsoralen) for acute graft-versus-host disease (GVHD within 100-days after HSCT). Photochemotherapy may be given as primary or later aGVHD therapy.

Exclusion Criteria:

* Patients with aGVHD after booster doses of stem-cells or donor-lymphocyte-infusions are not included.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with AML or ALL having received photochemotherapy for aGVHD evoked by HSCT given at Center for Allogeneic Stem Cell transplantation (CAST) between 1985 - end of 2004.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Graft-versus-leukemia (GVL) | 10-years after HSCT (2005 - 2015)
  i.e. abscence of relapse in malignant disease or minimal residual disease (MRD) i.e. threatening relapse in malignant disease demanding donor lymphocyte infusion (DLI).

SECONDARY OUTCOMES:
Death | 10-years after HSCT (2005 - 2015)
  Competing event
Retransplantation | 10-years after HSCT (2005 - 2015)
  Competing event
Donor Lymphocyte Infusion (DLI) | 10-years after HSCT (2005 - 2015)
  Competing event

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Feldreich, M.D., Principal Investigator — Division of Therapeutic Immunology, Department of Laboratory Medicine, Karolinska Institute; Olle Ringden, Professor, Study Director — Division of Therapeutic Immunology, Department of Laboratory Medicine, Karolinska Institute; Brigitta Omazic, PhD, Study Chair — Department of Oncology and Pathology,
Locations (1):
- Department of Dermatology, Karolinska University Hospital Huddinge, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Background] Thomas E, Storb R, Clift RA, Fefer A, Johnson FL, Neiman PE, Lerner KG, Glucksberg H, Buckner CD. Bone-marrow transplantation (first of two parts). N Engl J Med. 1975 Apr 17;292(16):832-43. doi: 10.1056/NEJM197504172921605. No abstract available. PMID 234595
- [Background] Ringden O, Witherspoon RP, Storb R, Ekelund E, Thomas ED. Increased in vitro B-cell IgG secretion during acute graft-versus-host disease and infection. Observations in 50 human marrow transplant recipients. Blood. 1980 Feb;55(2):179-86. PMID 6986176
- [Background] Ringden O, Sundberg B, Lonnqvist B, Tollemar J, Gahrton G, Nilsson B. Allogeneic bone marrow transplantation for leukemia: factors of importance for long-term survival and relapse. Bone Marrow Transplant. 1988 Jul;3(4):281-90. PMID 3048493
- [Background] Alyea EP, DeAngelo DJ, Moldrem J, Pagel JM, Przepiorka D, Sadelin M, Young JW, Giralt S, Bishop M, Riddell S. NCI First International Workshop on The Biology, Prevention and Treatment of Relapse after Allogeneic Hematopoietic Cell Transplantation: report from the committee on prevention of relapse following allogeneic cell transplantation for hematologic malignancies. Biol Blood Marrow Transplant. 2010 Aug;16(8):1037-69. doi: 10.1016/j.bbmt.2010.05.005. Epub 2010 May 24. PMID 20580849
- [Background] Horowitz MM, Gale RP, Sondel PM, Goldman JM, Kersey J, Kolb HJ, Rimm AA, Ringden O, Rozman C, Speck B, et al. Graft-versus-leukemia reactions after bone marrow transplantation. Blood. 1990 Feb 1;75(3):555-62. PMID 2297567
- [Background] Ringden O, Labopin M, Solders M, Beelen D, Arnold R, Ehninger G, Milpied N, Niederwieser D, Hamladji RM, Kyrcz-Krzemien S, Ganser A, Socie G, Stelljes M, Volin L, Craddock C, Mohty M; Acute Leukaemia Working Party of the European Group for Blood and Marrow Transplantation. Who is the best hematopoietic stem-cell donor for a male patient with acute leukemia? Transplantation. 2014 Sep 15;98(5):569-77. doi: 10.1097/TP.0000000000000102. PMID 24798307
- [Background] Strauss GH, Bridges BA, Greaves M, Hall-Smith P, Price M, Vella-Briffa D. Inhibition of delayed hypersensitivity reaction in skin (DNCB test) by 8-methoxypsoralen photochemotherapy. Possible basis for pseudo-promoting action in skin carcinogenesis? Lancet. 1980 Sep 13;2(8194):556-9. doi: 10.1016/s0140-6736(80)91992-3. PMID 6106738
- [Background] Wolf P, Nghiem DX, Walterscheid JP, Byrne S, Matsumura Y, Matsumura Y, Bucana C, Ananthaswamy HN, Ullrich SE. Platelet-activating factor is crucial in psoralen and ultraviolet A-induced immune suppression, inflammation, and apoptosis. Am J Pathol. 2006 Sep;169(3):795-805. doi: 10.2353/ajpath.2006.060079. PMID 16936256
- [Background] Glucksberg H, Storb R, Fefer A, Buckner CD, Neiman PE, Clift RA, Lerner KG, Thomas ED. Clinical manifestations of graft-versus-host disease in human recipients of marrow from HL-A-matched sibling donors. Transplantation. 1974 Oct;18(4):295-304. doi: 10.1097/00007890-197410000-00001. No abstract available. PMID 4153799
- [Background] Parrish JA, Fitzpatrick TB, Tanenbaum L, Pathak MA. Photochemotherapy of psoriasis with oral methoxsalen and longwave ultraviolet light. N Engl J Med. 1974 Dec 5;291(23):1207-11. doi: 10.1056/NEJM197412052912301. No abstract available. PMID 4422691
- [Background] Ringden O, Karlsson H, Olsson R, Omazic B, Uhlin M. The allogeneic graft-versus-cancer effect. Br J Haematol. 2009 Dec;147(5):614-33. doi: 10.1111/j.1365-2141.2009.07886.x. Epub 2009 Sep 4. PMID 19735262
- [Background] Hari P, Logan B, Drobyski WR. Temporal discordance between graft-versus-leukemia and graft-versus-host responses: a strategy for the separation of graft-versus-leukemia/graft-versus-host reactivity? Biol Blood Marrow Transplant. 2004 Nov;10(11):743-7. doi: 10.1016/j.bbmt.2004.07.006. PMID 15505605